CLINICAL TRIAL: NCT02676713
Title: Activating Blood, Dredging Liver and Nourishing Kidney Sequential Treatment for Endometriosis Associated Infertility - a Randomized Double-blind Placebo Controlled Study
Brief Title: Traditional Chinese Medicine Sequential Treatment for Endometriosis Associated Infertility
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Peking Union Medical College Hospital (Other); Beijing Hospital (Other Government); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other); The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Zhao RuiHua, Chief Physician, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GAMHospital; 2014BAI10B08 (Other Grant/Funding Number: 12th Five-Year National S&T Planed Project)
Record Dates: First submitted 2015-08-16; First posted 2016-02-08 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Endometriosis; Infertility
Keywords: Traditional Chinese Medicine; Chinese Herbal
MeSH Terms: conditions — Endometriosis; Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TCM Sequential Treatment (Experimental): After conservative surgery, patients start to take pre-ovulation decoction for 14 days. Each menstrual period 2～5 days, patients start to take pre-ovulation decoction. If ultrasonography found ovulation, change to take post-ovulation decoction. If having taken 14 days, ultrasonography found LUFS or no follicle develop maturity, change to take post-ovulation decoction. Taking post-ovulation decoction for 14 days, or continue to next time menstruation. Taking medication for six menstrual cycles.
  Pre-ovulation decoction is HuoXueXiaoYi decoction, and post-ovulation decoction is BuShenZhuYun decoction. 2 bags each time, 2 times a day, fused with hot water, 1 hour after dinner.
  All drugs are tcm formula granules, manufactured by Jiangyin Tianjiang Pharmaceutical Co. ltd
  Interventions: Drug: pre-ovulation Decoction; Drug: post-ovulation Decoction
- Placebo (Placebo Comparator): After conservative surgery, patients start to take pre-ovulation decoction(placebo) for 14 days. Each menstrual period 2～5 days, patients start to take pre-ovulation decoction. If ultrasonography found ovulation, change to take post-ovulation decoction. If having taken 14 days, ultrasonography found luteinized unruptured follicle syndrome (LUFS) or no follicle develop maturity, change to take post-ovulation decoction. Taking post-ovulation decoction(placebo) for 14 days, or continue to next time menstruation. Taking medication for six menstrual cycles. 2 bags each time, 2 times a day, fused with hot water, 1 hour after dinner.
  Pre-ovulation decoction and post-ovulation decoction is placebo, manufactured by Jiangyin Tianjiang Pharmaceutical Co. ltd
  Interventions: Drug: pre-ovulation Decoction(placebo); Drug: post-ovulation Decoction(placebo)

INTERVENTIONS:
Drug: pre-ovulation Decoction — HuoXueXiaoYi Decoction(Bupleurum 10g, Cyperus 10g, Salvia miltiorrhiza 20g, Red peony 10g,etc)has activating blood and absorbing clots effect, can inhibit the growth of ectopic endometrium, promote follicular growth, maturity, improve ovulation and the receptivity of endometrium.
  Other Names: HuoXueXiaoYi Decoction
  Arms: TCM Sequential Treatment
Drug: post-ovulation Decoction — BuShenZhuYun Decoction(Bupleurum 10g,Poria 15g, Atractylodes 15g,Ligustrum 15g,etc) has dredging liver and nourishing kidney effect, can improve the function of corpus luteum.
  All are made into granules.
  Other Names: BuShenZhuYun Decoction
  Arms: TCM Sequential Treatment
Drug: pre-ovulation Decoction(placebo) — Composition of maltodextrin, lactose, edible pigment, taste masking agent.
  Other Names: placebo
  Arms: Placebo
Drug: post-ovulation Decoction(placebo) — Composition of maltodextrin, lactose, edible pigment, taste masking agent.
  Other Names: placebo
  Arms: Placebo

SUMMARY:
Endometriosis is a common, chronic disease. 30% to 50% of women with endometriosis are infertile. There is moderate quality evidence that laparoscopic surgery to treat mild and moderate endometriosis increases live birth or ongoing pregnancy rates. There was no evidence of benefit for post-surgical hormonal suppression of endometriosis compared to surgery alone for the outcomes of pregnancy rates. Past studies have confirmed that Chinese herbal medicine can inhibit post-surgical endometriosis recurrence, increase pregnancy rate.This study evaluates the efficacy and safety of Traditional Chinese Medicine Sequential Treatment of endometriosis-associated infertility. The study objective is to confirm that clinical pregnancy rate of patients with endometriosis-associated infertility post-conservative surgery accepting Chinese medicine activating blood, dredging liver and nourishing kidney sequential treatment is higher than expectant treatment.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, multicenter, prospective clinical study, conducted in China (six research centers).

204 cases of patients with endometriosis-associated infertility confined with Syndrome of qi stagnation blood stasis pattern in TCM after conservative surgery will be recruited. Patients will be randomly divided into two groups: experimental group (TCM Sequential Treatment) and control group (placebo). All the patients are treated for six menstrual cycles, taking pre-ovulation decoction before ovulation and post-ovulation decoction after ovulation. Pre-ovulation decoction of experimental group is HuoXueXiaoYi decoction, and post-ovulation decoction is BuShenZhuYun decoction. The drug of control group is placebo.

Each menstrual cycle, patient is monitored of antral follicle count (AFC), ovulation, endometrial thickness, and endometrial blood flow by ultrasonography, and need fill TCM syndrome rating scale, pictorial blood loss assessment chart (PBAC), and the visual analogue scale(VAS).The 1st, 3rd, 6th menstrual cycle after surgery, the level of serum female hormone (FSH, LH, E2) are detected in menstrual period of 2 to 5 days, and female hormone (E2, P) in the middle of the corpus luteum 6-9 days.

Patient must be security check (blood routine, urine routine, liver and kidney function, electrocardiogram) before and after drug treatment. Such as patients find pregnancy during medication, adopt the security check in finding pregnancy 7 days.

Patients after amenorrhea need to be confirmed pregnancy by serum β-HCG detection. According to the level of serum HCG, E2 and P and clinical symptoms, corresponding tocolytic treatment will be given. At 6～8 weeks of pregnancy, patient need to be confirmed the clinical pregnancy by ultrasonography. If confirmed the clinical pregnancy (at least having one heart throb in intrauterine gestational sac), patient need to be confirmed ongoing pregnancy by ultrasonography at the 12～14 weeks of pregnancy.

In the process of the entire study, adverse events will be closely observed, and the frequency and severity of adverse events will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of endometriosis, infertility, with Syndrome of qi stagnation blood stasis pattern in TCM ;
2. The first time undergoing Laparoscopic or laparoscopy combined surgery , in lined with endometriosis-related infertility, tubal patency or obstruction lightly;
3. EFI score greater than 4 points;
4. Early follicular phase FSH≤10mIU / L;
5. 28 days of the menstrual cycle ± 7 days;
6. Female patients between 20-35 years old;
7. No previous history of severe drug allergies;
8. Past Three-month no taking hormone drugs such as danazol, Gestrinone, GnRHa;
9. No severe primary brain vascular diseases, liver, kidney and hematopoietic systems diseases, no history of mental illness, no drugs, alcohol, tobacco, caffeine dependent history;
10. Have signed informed consent

Exclusion Criteria:

1. Associated with uterine fibroids, the diameter greater than 4cm, adenomyosis, pelvic tuberculosis, endometrial tuberculosis, intrauterine adhesions, polycystic ovary syndrome, hyperprolactinemia, thyroid dysfunction patients.
2. Serious history of drug allergy.
3. Male factor infertility.
4. The couple separated persons.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 204 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-05 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate | six menstrual cycles（each cycle is 28±7 days）
  Pregnancy rate is defined as the proportion of participants finding pregnancy after amenorrhea and confirming serumβ-HCG positive.

SECONDARY OUTCOMES:
Clinical pregnancy rate (with intrauterine pregnancy sac) | at 6～8 weeks of pregnancy
  defined as the proportion of participants confirmed there are at least one gestational sac in uterine cavity (No matter whether there is a heart throb) by ultrasonography.
Clinical pregnancy rate (with a heart throb) | at 6～8 weeks of pregnancy
  defined as the proportion of participants confirmed at least having one heart throb in intrauterine gestational sac by ultrasonography.
Continued pregnancy rate | at the 12～14 weeks of pregnancy
  defined as the proportion of participants confirmed at least one live fetuses by ultrasonography.

OTHER OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events | six menstrual cycles（each cycle is 28±7 days）
  Treatment-emergent Adverse Events were assessed by CTCAE v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Zhao, Doctor, Study Chair — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (6):
- China (6):
  - The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine, Hefei, Anhui
  - Beijing Obstetrics and Gynecology Hospital,Captial Medical University, Beijing, Beijing Municipality
  - GAMHospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou University of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Traditional Chinese Medicine Hospital of Guangdong Province, Guangzhou, Guangdong
  - Beijng Hospital, Beijng

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duffy JM, Arambage K, Correa FJ, Olive D, Farquhar C, Garry R, Barlow DH, Jacobson TZ. Laparoscopic surgery for endometriosis. Cochrane Database Syst Rev. 2014 Apr 3;(4):CD011031. doi: 10.1002/14651858.CD011031.pub2. PMID 24696265
- [Background] Yap C, Furness S, Farquhar C. Pre and post operative medical therapy for endometriosis surgery. Cochrane Database Syst Rev. 2004;2004(3):CD003678. doi: 10.1002/14651858.CD003678.pub2. PMID 15266496
- [Result] Zhao RH, Hao ZP, Zhang Y, Lian FM, Sun WW, Liu Y, Wang R, Long L, Cheng L, Ding YF, Song DR, Meng QW, Wang AM. Controlling the recurrence of pelvic endometriosis after a conservative operation: comparison between Chinese herbal medicine and western medicine. Chin J Integr Med. 2013 Nov;19(11):820-5. doi: 10.1007/s11655-012-1247-z. Epub 2012 Dec 22. PMID 23292545
- [Derived] Zhao RH, Liu Y, Lu D, Wu Y, Wang XY, Li WL, Zeng C, Meng QW, Lian FM, Zhou J, Shi Y, Sun WW, Han Q, Tang Y, Shi G. Chinese Medicine Sequential Therapy Improves Pregnancy Outcomes after Surgery for Endometriosis-Associated Infertility: A Multicenter Randomized Double-blind Placebo Parallel Controlled Clinical Trial. Chin J Integr Med. 2020 Feb;26(2):92-99. doi: 10.1007/s11655-019-3208-2. Epub 2020 Jan 29. PMID 31997236